CLINICAL TRIAL: NCT03050190
Title: A Phase I/II Multiple Center Trial of 4SCAR19 Cells in the Treatment of Relapsed and Refractory B Cell Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-16001
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: B-cell Malignancies
Keywords: CART therapy; 4SCAR19; CD19; B cell leukemia; B-ALL
MeSH Terms: conditions — Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic 4SCAR19 cells (Experimental): Patients who have relapsed and refractory B cell leukemia after chemotherapy will be treated prophylactically with CD19-specific gene-engineered T cells.
  Interventions: Genetic: Therapeutic 4SCAR19 cells

INTERVENTIONS:
Genetic: Therapeutic 4SCAR19 cells — Autologous 4th generation withdrawal lentiviral-transduced 4S CAR-T19

SUMMARY:
The study will evaluate safety and efficacy of a 4th generation chimeric antigen receptor gene-modified T cells targeting CD19 (4SCAR19) for patients with B cell malignancies. Clinical response and development of a standardized lentiviral vector and cell production protocol will be investigated. This is a phase I/II trial enrolling patients from multiple clinical centers.

DETAILED DESCRIPTION:
Background:

T cells modified with lentiviral chimeric antigen receptor (CAR) gene have been studied in different clinical settings. Recent successes suggest that increased costimulatory signaling in the CAR design is critical for long term efficacy. Activation of T cell response from large tumor burden may induce a severe response. To increase safety, a novel design using an inducible caspase 9 fusion gene has been incorporated in the CAR gene. A 4th generation CAR lentiviral vector (4SCAR) carrying T cell costimulatory signals for CD28/CD27 plus an inducible apoptotic caspase 9 gene has been established. The study aims to evaluate the activities of a new CAR gene-modified T cells targeting CD19-positive tumors based on a CD19-specific single chain gene constructed 4SCAR (4SCAR19).

Objective:

To evaluate safety and efficacy of administrating 4SCAR19 T cells to patients with CD19 positive B cell malignancies following a cyclophosphamide/fludarabine based conditioning regimen.

Eligibility:

Patients older than 6-month-old with CD19 positive B cells malignancies that have recurred after or refractory to standard therapy and is deemed incurable using standard treatment.

Design:

Participants will be screened based on cancer cell phenotype analyzed using flow cytometry or immunohistochemical staining methods.

Peripheral blood mononuclear cells (PBMC) will be obtained through apheresis, and T cells will be activated and modified to express the 4SCAR19 gene.

On Day -5 to -7, PBMC will be activated and enriched for T cells, which will be followed by 4SCAR19 lentiviral transduction. The total cell preparation time is approximately 5-7 days.

Participants will receive a preparative conditioning regimen comprising cyclophosphamide/fludarabine to prepare their immune system to accommodate the modified CAR T cells. The preparative regimen will be based on patient immune condition and consistent with standard chemotherapy conditioning regimen.

Participants will receive an infusion of the modified 4SCAR19 T cells and closely followed up for treatment-related responses.

Participants will be continuously monitored for CAR T cells and clinical responses at present timeline.

ELIGIBILITY:
Inclusion Criteria:

1. aged more than 6 months.
2. malignant B cell surface expression CD19 molecules.
3. the KPS score over 80 points, and survival time is more than 3 months.
4. greater Hgb 80 g/L.
5. no contraindications to solid and cell separation

Exclusion Criteria:

1. accompanied with other active diseases, the treatment is difficult to correct.
2. bacteria, fungus, or virus infection, unable to control.
3. people living with HIV.
4. active HBV and HCV infection.
5. of pregnancy and nursing mothers.
6. before entering the test of the use of glucocorticoid systemic treatment within a week.
7. confirmed before used CAR - but invalid

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of fourth generation anti CD19 CAR-T cells in patients with relapsed B cell malignancies using CTCAE 4 standard to evaluate the level of adverse events | 24 weeks
  physiological parameter (for safety, measuring cytokine response, fever, symptoms)

SECONDARY OUTCOMES:
Anti tumor activity of fourth generation anti CD19 CAR-T cells in patients with relapsed or refractory B cell malignancies | 1 year
  scale of CAR copies and leukemic cell burden (for efficacy)

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (2):
- China (2):
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - The First People's Hospital of Yunnan, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nair S, Wang JB, Tsao ST, Liu Y, Zhu W, Slayton WB, Moreb JS, Dong L, Chang LJ. Functional Improvement of Chimeric Antigen Receptor Through Intrinsic Interleukin-15Ralpha Signaling. Curr Gene Ther. 2019;19(1):40-53. doi: 10.2174/1566523218666181116093857. PMID 30444200